CLINICAL TRIAL: NCT02535767
Title: Determining a Tolerable Dose of Primaquine in G6PD-deficient Persons Without Malaria in Mali
Acronym: PQSAFETY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); Radboud University Medical Center (Other); University of Mississippi Medical Center (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-14495
Record Dates: First submitted 2015-08-07; First posted 2015-08-31 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Malaria
Keywords: Primaquine
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A: 0.40 mg/kg PQ G6PDd (Experimental): 0.40 mg/kg of primaquine (as a single dose) in G6PD-deficient individuals
  Interventions: Drug: Primaquine
- B: PQ in G6PDd (Experimental): A single dose of primaquine in G6PD-deficient men, exact dose to be decided by DSMB based on findings in previous dose group. The minimum change in dose from the last study dose is 0.05 mg/kg, and the maximum change is 0.20 mg/kg of primaquine). Dose is not to exceed 0.75 mg/kg primaquine.
  Interventions: Drug: Primaquine
- C: PQ in G6PDd (Experimental): A single dose of primaquine in G6PD-deficient men, exact dose to be decided by DSMB based on findings in previous dose group. The minimum change in dose from the last study dose is 0.05 mg/kg, and the maximum change is 0.20 mg/kg of primaquine). Dose is not to exceed 0.75 mg/kg primaquine.
  Interventions: Drug: Primaquine
- D: PQ G6PDn (Experimental): A single dose of primaquine in G6PD-normal men, at the highest tolerable dose determined by the DSMB, from previous dose groups.
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — A single low dose of primaquine will be crushed and dissolved in water, and administered in weight-based doses.

SUMMARY:
The purpose of this study is to determine the highest tolerable dose of primaquine within 0.75 mg/kg. A tolerable dose is defined as one in which:

* Two or fewer participants (< 30%) experience hemolysis;
* No participant experiences a drug-related serious adverse event; and
* No participant requires a blood transfusion.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to determine the highest tolerable dose of primaquine within 0.75 mg/kg. A tolerable dose is defined as one in which:

* Two or fewer participants (< 30%) experience hemolysis;
* No participant experiences a drug-related serious adverse event; and
* No participant requires a blood transfusion.

Design:

* This is an open-label, phase 2, dose-adjustment study.
* The initial primaquine dose will be 0.40 mg/kg. Subsequent dose groups will be selected depending on the occurrence of adverse events in the previous dose group. Once the highest tolerable dose in G6PD-deficient (G6PDd) individuals is established, a control group of G6PD normal malaria-free men will be enrolled and evaluated under the highest tolerable dose of primaquine.

Study Population:

* Malian men aged 18-50 years without malaria infection.
* The majority of study participants will be G6PDd.

Study Size: This study will enroll 7 participants per dose group. If all dose groups are tested, this study will enroll approximately 28 participants.

Study visit and duration:

* Each participant will be followed for 28 days.
* Participants will be evaluated for hemolysis and adverse events on Days 1-10, 14, and 28 following their assigned primaquine dose.

Primary objective:

To measure the change in hemoglobin among G6PD deficient west-African men following a single low-dose of primaquine not to exceed 0.75 mg/kg.

Secondary objectives:

1. To measure the occurrence of adverse events, graded by severity, at each primaquine dose among G6PD deficient men
2. To measure the occurrence of markers of acute hemolytic anemia (AHA), at each primaquine dose among G6PD deficient men. AHA markers will include:

   * Absolute and fractional change in hemoglobin on day 7 vs. baseline
   * Urine color
   * Reticulocyte count
   * Bilirubin (both total and direct)
   * Methemoglobin concentration
   * Development of physical signs or symptoms of hemolytic anemia
3. To compare the change in hemoglobin, frequency and severity of adverse events, and occurrence of markers of AHA between G6PD deficient and non-deficient participants receiving the highest tolerable primaquine dose
4. To measure G6PD enzyme activity (semiquantitative testing, U / gHb)
5. To measure the pharmacokinetics of primaquine, carboxyprimaquine, and other metabolites according to plasma concentrations.
6. To genotype participant blood samples for cytochrome P450 2D6 (CYP2D6) single nucleotide polymorphisms (SNPs), to determine if potential hemolysis in G6PDd individuals is affected by CYP2D6 metabolizer status (e.g. weak metabolizers and/or intermediate metabolizers)

ELIGIBILITY:
Inclusion Criteria:

* Males ages 18- 50 (inclusive)
* Ability to swallow oral medication
* Informed consent
* Willing and able to participate in the study for 28 days

For the G6PDd participants:

* G6PDd defined by Carestart 3 rapid diagnostic test or
* The OSMMR2000 G6PD qualitative test

For the G6PDn participants:

* G6PDn defined by Carestart 3 rapid diagnostic test or
* The OSMMR2000 G6PD qualitative test

Exclusion Criteria:

* Moderate to severe anemia (Hb < 10 g/dL)
* Malaria infection by blood smear
* Individuals with known positive HIV test
* Individuals with known positive hepatitis B test.
* Known allergy to study drugs
* Current use of medication (for tuberculosis, HIV, or any drugs that have hemolytic potential in G6PDd individuals including sulphonamides, dapsone, nitrofurantoin, nalidixic acid, ciprofloxacin, methylene blue, toluidine blue, phenazopyridine, and co-trimoxazole)
* The individual is unwilling to abstain from the ingestion of grapefruit-containing products from 72 hours prior to the start of dosing until the study is complete
* Use of antimalarials within 2 weeks before contact with the study team as reported by the patient
* History of blood transfusion or a bleed of > 500 mLs within the last 3 months, as reported by the patient
* Reported history of high alcohol intake (> 14 units per week, each unit is equivalent to 10 g of alcohol (1 glass of wine or 1 bottle of beer or one shot of distilled spirits), within 6 months of study as reported by the patient
* Reported use of illicit drugs (marijuana, heroin, cocaine, methamphetamine) or dependence within 6 months of study, as reported by the patient
* Participants who vomit within 1 hour after administration of primaquine (will be removed from the analysis and will not count towards the total sample size, though they will be followed as any other enrolled individual)
* Already enrolled in this study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Primary outcome: the change in hemoglobin concentration from baseline levels following a single low-dose of primaquine not to exceed 0.75 mg/kg. | Between day 0 and day 10.

SECONDARY OUTCOMES:
To measure the occurrence of adverse events, graded by severity, at each primaquine dose among G6PD deficient men | Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 14, and 28
  Severity:
  1. = mild
  2. = moderate
  3. = severe
  4. = life threatening
To measure the occurrence of absolute and fractional change in hemoglobin concentration (g/dL) on day 7 vs. baseline at each primaquine dose among G6PD deficient men, in comparison with G6PD normal men | Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 14, and 28
To measure the occurrence of reticulocytosis (by microscopic quantification of reticulocytes stained with brilliant cresyl blue / 1,000 RBCs) on each day of followup, at each primaquine dose, among G6PD deficient men, in comparison with G6PD normal men | Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 14, and 28
To monitor methemoglobin levels (%) on each day of followup, at each primaquine dose among G6PD deficient men, in comparison with G6PD normal men | Days 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 14, and 28
  Use of a Masimo Rad-57 pulse oximeter that measures methemoglobin levels non-invasively, based on absorption of light through the fingertip.
To determine G6PD enzyme activity (semiquantitative testing, U/g Hb) | Day 0
  Semiquantitative testing will be performed on frozen blood samples to determine G6PD activity on day of enrolment
Area Under Curve (AUC) for primaquine | Hours 1, 2, 4, 6, 8, and 24 after primaquine administration
  Pharmacokinetic analysis of plasma concentration of primaquine at all sampled timepoints
Maximal concentration (Cmax) for primaquine | Hours 1, 2, 4, 6, 8, and 24 after primaquine administration
  Pharmacokinetic analysis of plasma concentration of primaquine at all sampled timepoints
Area Under Curve (AUC) for carboxyprimaquine | Hours 1, 2, 4, 6, 8, and 24 after primaquine administration
  Pharmacokinetic analysis of plasma concentration of carboxyprimaquine
Maximal concentration (Cmax) for carboxyprimaquine | Hours 1, 2, 4, 6, 8, and 24 after primaquine administration
  Pharmacokinetic analysis of plasma concentration of carboxyprimaquine
Area Under Curve (AUC) for select minor metabolites of primaquine | Hours 1, 2, 4, 6, 8, and 24 after primaquine administration
  Pharmacokinetic analysis of plasma concentration of metabolites of primaquine, exact metabolites to be determined by ongoing in vivo studies (including 5-hydroxyprimaquine)
Maximal concentration (Cmax) for select minor metabolites of primaquine | Hours 1, 2, 4, 6, 8, and 24 after primaquine administration
  Pharmacokinetic analysis of plasma concentration of metabolites of primaquine, exact metabolites to be determined by ongoing in vivo studies (including 5-hydroxyprimaquine)
Cytochrome P450 (CYP) 2D6 genotyping | Day 0
  To determine whether a correlation between CYP 2D6 metabolism (weak metabolizer, intermediate metabolizer, normal metabolizer, ultrarapid metabolizer) and hemolysis exists.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Gosling, PhD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- Malaria Research and Training Centre, Bamako, Mali

REFERENCES:
- [Derived] Chotsiri P, Mahamar A, Diawara H, Fasinu PS, Diarra K, Sanogo K, Bousema T, Walker LA, Brown JM, Dicko A, Gosling R, Chen I, Tarning J. Population pharmacokinetics of primaquine and its metabolites in African males. Malar J. 2024 May 21;23(1):159. doi: 10.1186/s12936-024-04979-y. PMID 38773528
- [Derived] Chen I, Diawara H, Mahamar A, Sanogo K, Keita S, Kone D, Diarra K, Djimde M, Keita M, Brown J, Roh ME, Hwang J, Pett H, Murphy M, Niemi M, Greenhouse B, Bousema T, Gosling R, Dicko A. Safety of Single-Dose Primaquine in G6PD-Deficient and G6PD-Normal Males in Mali Without Malaria: An Open-Label, Phase 1, Dose-Adjustment Trial. J Infect Dis. 2018 Mar 28;217(8):1298-1308. doi: 10.1093/infdis/jiy014. PMID 29342267